CLINICAL TRIAL: NCT04807244
Title: Randomized-controlled and Non-controlled Intervention Trial: Treatment of Deep Carious Lesions in Permanent Molars
Brief Title: Treatment of Deep Carious Lesions With Selective Caries Removal, Partial or Full Pulpotomy
Acronym: Vitapulp
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Septodont (Industry); 3M (Industry)
Responsible Party: Principal Investigator, Falk Schwendicke, Head of the Department for Oral Diagnostics, Digital Health and Health Services Research, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EA4/249/20
Record Dates: First submitted 2021-03-11; First posted 2021-03-19 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Irreversible Pulpitis; Reversible Pulpitis; Dentine Caries
Keywords: Partial Pulpotomy; Full Pulpotomy; Selective Caries Removal
MeSH Terms: interventions — tricalcium silicate

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial and Prospective Non-controlled Intervention Trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Every patient has to give informed consent for participating in one of both study arms. To avoid clustering, only one tooth per patient can be included. Arm A is designed as a randomized-controlled and arm B as a non-controlled intervention trial.
  The intervention in study arm B will be conducted adapted to the clinical findings after entering slightly the pulp chamber. Depending on the pulpal bleeding time, either a partial pulpotomy or a full pulpotomy will be conducted, according to the predefined protocol mentioned in "treatment protocol for arm A". Due to the experimental design, only single blinding of the patient is feasible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment of deep carious lesions: Randomized-controlled trail (Other): Teeth with reversible pulpitis will be included accordingly to the inclusion criteria (see below). After randomization, teeth will be treated either with selective caries removal (indirect pulp capping) or partial pulpotomy pursuant to the below described clinical protocol. The intention of this study arm is to evaluate both therapies.
  Interventions: Procedure: Selective Caries Removal with Biodentine™; Procedure: Partial Pulpotomy with Biodentine™; Procedure: Direct composite filling after selective caries removal/full pulpotomy/partial pulpotomy
- Treatment of deep carious lesions: Prospective non-controlled intervention trial (Other): Teeth with reversible pulpitis according to the inclusion criteria (see below) will be included. Depending on the clinical situation, a partial or full pulpotomy will be conducted accordingly to the defined clinical protocols (see below). In this study arm, we want to evaluate 1) different times of pulpal bleeding before pulp capping and 2) partial versus full pulpotomy on the clinical outcome in teeth with irreversible pulpitis.
  Interventions: Procedure: Full Pulpotomy with Biodentine™; Procedure: Direct composite filling after selective caries removal/full pulpotomy/partial pulpotomy

INTERVENTIONS:
Procedure: Selective Caries Removal with Biodentine™ — 1. Rubber dam placement
  2. Cleaning of the tooth and rubber dam with ethanol 98%
  3. Caries removal: Removal of protruding parts of enamel/dentin with high-speed round bur with continuous water cooling, caries removal with a low-speed round bur; peripheral caries is removed until only hard dentin is left, while the pulp wall is excavated until reaching leathery dentin
  4. Disinfection of the leathery dentin 5 ml 1% NaOCl (speed: 1 ml per min)
  5. Indirect pulp capping (layer of 1-2 mm) of the carious lesion with Biodentine™ (15 min setting time after mixing)
  Arms: Treatment of deep carious lesions: Randomized-controlled trail
Procedure: Partial Pulpotomy with Biodentine™ — 1. Rubber dam placement
  2. Cleaning of the tooth and rubber dam with ethanol 98%
  3. Caries removal: Removal of protruding parts of enamel/dentin with high-speed round bur with continuous water cooling, caries removal with a low-speed round bur; before accessing the pulp chamber, the central caries will be left, peripheral caries will be excavated completely
  4. Disinfection of the leathery dentin 5 ml NaOCl 1% (speed: 1 ml per min)
  5. Accessing the pulp chamber with a high-speed round bur and removal of 2-3 mm pulp tissue; irrigation with 2 ml NaOCl 1%
  6. Hemostasis will be achieved with a sterile foam pellet soaked with NaOCl 1% with gentle pressure to the pulp for 3 min
  7. If hemostasis could not be achieved within 3 min, step 6 will be repeated once. In case of no hemostasis, transfer of the case to Intervention: "full pulpotomy with Biodentine"
  8. Confirmed hemostasis: pulp capping with Biodentine™ (layer min. 2-3 mm, 15 min setting time after mixing)
  Arms: Treatment of deep carious lesions: Randomized-controlled trail
Procedure: Full Pulpotomy with Biodentine™ — 1. Rubber dam placement
  2. Cleaning of the tooth and rubber dam with ethanol 98%
  3. Caries removal: Removal of protruding parts of enamel/dentin with high-speed round bur with continuous water cooling, caries removal with a low-speed round bur; before accessing the pulp chamber, the central caries will be left, peripheral caries will be excavated completely
  4. Disinfection of the leathery dentin 5 ml NaOCl 1% (speed: 1 ml per min)
  5. Accessing the pulp chamber with a high-speed round bur and removal of the entire pulp chamber roof; full pulpotomy to stump level with a high-speed round bur under continuous irrigation with 5 ml NaOCl 1%
  6. Hemostasis will be achieved with a sterile foam pellet soaked with NaOCl 1% with gentle pressure to the pulp for 3 min
  7. If hemostasis could not be achieved within 3 min, step 6 will be repeated once. In case of no hemostasis, exclusion.
  8. Confirmed hemostasis: pulp capping with Biodentine™ (layer min. 2-3 mm, 15 min setting time after mixing)
  Arms: Treatment of deep carious lesions: Prospective non-controlled intervention trial
Procedure: Direct composite filling after selective caries removal/full pulpotomy/partial pulpotomy — 1. Dentin cleaning with a low-speed round bur
  2. Use of Scotchbond Universal™ and Filtek Supreme XTE™ according to manufacturer's recommendation

SUMMARY:
The optimal treatment of deep caries lesions extended to the inner third of dentin is still under discussion. Cariologists prefer selective caries removal, meanwhile endodontists recommend partial pulpotomy. So far, no clinical trial compared both interventions against each other. Additionally, current literature indicates alternative treatment options for irreversible pulpitis besides conventional orthograde root canal treatments like the partial or full pulpotomy. Existing clinical studies on this topic were using different clinical protocols, especially with regards to the accepted time to achieve hemostasis. It is still unclear, if the pulpal bleeding time prior to the capping procedure affects the outcome of partial or full pulpotomy.

DETAILED DESCRIPTION:
Goals of the study

In consequence, the investigators aim to proof the effectiveness of different therapies and protocols in two study arms, depending on the initial diagnosis:

Arm A: Randomized-controlled clinical non-inferiority trial:

Teeth with reversible pulpitis will be included accordingly to the inclusion criteria (see below). After randomization, teeth will be treated either with selective caries removal (indirect pulp capping) or partial pulpotomy pursuant to the below described clinical protocol. The intention of this study arm is to evaluate both therapies.

Arm B: Prospective non-controlled clinical intervention trial

Teeth with reversible pulpitis according to the inclusion criteria (see below) will be included. Depending on the clinical situation, a partial or full pulpotomy will be conducted accordingly to the defined clinical protocols (see below). In this study arm, the investigators want to evaluate 1) different times of pulpal bleeding before pulp capping and 2) partial versus full pulpotomy on the clinical outcome in teeth with irreversible pulpitis.

Primary hypothesis:

There is no statistically significant difference in the clinical success (absence of any clinical symptoms and signs of inflammation) between both treatments.

Secondary hypothesis:

There is no statistically significant difference in the radiographical success (absence of any pathosis) between both treatments.

Duration of the study:

The study is estimated to complete enrollment within 18 months from study initiation. In cases of unforeseeable events, enrollment will remain open until the study goal is met. For each subject, participation will be a maximum of three years.

Products intended use

All products the investigators intend to use are registered medicine products and well established on the market:

• Biodentine™ (Septodont, Saint-Maur-des-Fossés, France): Biodentine™ is a hydraulic calcium silicate cement (HSC), which is commonly used for vital pulp therapy in both, children and adults. Many clinical trials were successfully conducted with this material. Compared to other HSC, the effect of tooth staining is much less likely and the clinical perfomance is comparable to other HSC. The main advantage of Biodentine™ compared to other HSC is, that Biodentine™ needs only 15 min for setting up, other HSC show significantly longer settings times. Septodont recommends using a self-etch adhesive in combination with Biodentine™.

• Scotchbond Universal™ and Filtek Supreme XTE™ Scotchbond Universal™ is a self-etch adhesive and Filtek Supreme XTE™ is a universal restorative material for direct restorations (3M, Saint Paul, Minnesota, USA). Both materials are commercially available since many years and approved in several clinical trials.

Product acquisition

Biodentine™, Scotchbond Universal™ and Filtek Supreme XTE™ will be sponsored by the manufacturer. All other materials of routine use will be purchased by the centers.

Potential benefits and risks to patients

Every effort is taken during all treatments to minimize the risks to the patients. The primary goal of arms A and B is to evaluate three well established interventions. In consequence, the investigators expect no higher risks to the patients compared to routine treatments in our clinic.

The benefit in participating for the patient is, that the investigators offer minimally invasive interventions for lower costs than usual. In cases of failure, the investigators follow our protocol as described in "failure management".

Methods:

Study design:

Single-blind multi-center study with two arms involving two hundred and forty-nine (249) subjects undergoing a deep caries therapy. Four dental clinics with board certified endodontists contribute to this study in terms of patient recruitment and treatment. The centers are:

1. Charité - Universitätsmedizin Berlin, Department for Oral Diagnostics, Digital Health and Health Services Research, Aßmannshauser Str. 4-6, 14197 Berlin Local principal investigator and study leader: Dr. Sascha Herbst
2. B1 Zahnärzte, Clayallee 177, 14195 Berlin Local principal investigator: Dr. Claus Schüttler-Janikulla
3. Endo Berlin Süd, Alt-Buckow 9-11, 12349 Berlin Local principal investigator: ZÄ Olga Bleckmann
4. Dentalsplace, Kurfürstendamm 22 Local principal investigator: Dr. Markus Lietzau, M.Sc.

Every patient has to give informed consent for participating in one of both study arms. To avoid clustering, only one tooth per patient can be included. Arm A is designed as a randomized-controlled and arm B as a non-controlled intervention trial.

The intervention in study arm B will be conducted adapted to the clinical findings after entering slightly the pulp chamber. Depending on the pulpal bleeding time, either a partial pulpotomy or a full pulpotomy will be conducted, according to the predefined protocol mentioned in "treatment protocol for arm A". Due to the experimental design, only single blinding of the patient is feasible.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 a Health status
* No contributory systemic diseases with influence to the immune system or coagulation system

Tooth-related factors

* Type: Permanent molars
* Mature roots
* Caries extended to >2/3 of dentin and expected pulp exposure performing non-selective caries removal (Only study arm "partial pulpotomy": Pulp exposure after non-selective caries removal)
* Sensibility: +/++; prolonged <5s
* Pain only on stimulus (hot/cold) and not prolonged or no pain
* No tenderness to palpation
* No tenderness to percussion
* Periodontal probing depth <4 mm
* No pathologic tooth mobility
* No swelling
* No fistula
* No swelling
* Radiograph: Periapical status with physiological appearance (PAI Score I or II)
* No partial/full crown restauration
* Tooth has to be restorable
* Pulpal diagnosis reversible pulpitis

Exclusion Criteria:

* Age < 18 a
* Health status with above mentioned contributory diseases (immunosuppression, or diseases related to the coagulation system)
* Deciduous teeth
* Immature roots
* Caries extending less than <2/3 of dentin
* (Only study arm "partial pulpotomy": No pulp exposure after non-selective caries removal)
* Tooth sensibility +++ or prolonged > 5 s
* Severe pain, prolonged on stimulus (hot/cold), dull, throbbing, spontaneous pain
* Tenderness to palpation +
* Periodontal probing depth >3 mm
* Tooth mobility grade >Score I
* Swelling present
* Fistula present
* Radiograph: Apical periodontitis or apical rarefaction
* Partial or full crown restauration in situ
* Tooth is non-restorable
* Diagnosis: Irreversible pulpitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 249 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients with positive reaction to cold testing | 36 months
  Tooth sensibility with endo coldspray (-40°C) (positive or negative reaction of the patient)
Number of patients without mobile teeth | 36 months
  Tooth mobility testing with two fingers according to the tooth mobility score (0-III)
Number of patients with negative reaction to palpation testing | 36 months
  Palpation testing with a finger and little pressure (tenderness to palpation or no tenderness to palpation)
Number of patients with negative reaction to percussion testing | 36 months
  Percussion testing of the treated tooth: backside of dental mirror (tenderness to percussion or no tenderness to percussion)
Number of patients with periodontal probing depths within normal limits | 36 months
  Probing depths with a periodontal probe in mm
Number of Patients without clinical signs of inflammation | 36 months
  Screening the oral mucosa for swelling, fistula and erythema

SECONDARY OUTCOMES:
Number of patients with a PAI score of I - II | 36 months
  Evaluation of the periapical status on periapical radiographs via periapical index (PAI)

CONTACTS AND LOCATIONS:
Overall Officials: Falk Schwendicke, Prof., Study Director — Charite University, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adl A, Javanmardi S, Abbaszadegan A. Assessment of tooth discoloration induced by biodentine and white mineral trioxide aggregate in the presence of blood. J Conserv Dent. 2019 Mar-Apr;22(2):164-168. doi: 10.4103/JCD.JCD_466_18. PMID 31142987
- [Background] Awawdeh L, Al-Qudah A, Hamouri H, Chakra RJ. Outcomes of Vital Pulp Therapy Using Mineral Trioxide Aggregate or Biodentine: A Prospective Randomized Clinical Trial. J Endod. 2018 Nov;44(11):1603-1609. doi: 10.1016/j.joen.2018.08.004. Epub 2018 Oct 3. PMID 30292451
- [Background] Duncan HF, Bjorndal L, van der Sluis L, Rechenberg DK, Simon S, Cooper PR, Ricucci D, Galler K. Third European Society of Endodontology (ESE) research meeting: ACTA, Amsterdam, The Netherlands, 26th October 2018: Deep caries and the exposed pulp: current and emerging therapeutic perspectives. Int Endod J. 2019 Feb;52(2):135-138. doi: 10.1111/iej.13059. No abstract available. PMID 30644590
- [Background] Burke FJT, Crisp RJ, Cowan AJ, Raybould L, Redfearn P, Sands P, Thompson O, Ravaghi V. A Randomised Controlled Trial of a Universal Bonding Agent at Three Years: Self Etch vs Total Etch. Eur J Prosthodont Restor Dent. 2017 Dec 1;25(4):220-227. doi: 10.1922/EJPRD_01692Burke08. PMID 29182212
- [Background] Camilieri J (2015) Mineral trioxide aggregate: present and future developments Endodontic Topics Volume 31, 31-46.
- [Background] de Paris Matos T, Perdigao J, de Paula E, Coppla F, Hass V, Scheffer RF, Reis A, Loguercio AD. Five-year clinical evaluation of a universal adhesive: A randomized double-blind trial. Dent Mater. 2020 Nov;36(11):1474-1485. doi: 10.1016/j.dental.2020.08.007. Epub 2020 Sep 12. PMID 32933775
- [Background] Galani M, Tewari S, Sangwan P, Mittal S, Kumar V, Duhan J. Comparative Evaluation of Postoperative Pain and Success Rate after Pulpotomy and Root Canal Treatment in Cariously Exposed Mature Permanent Molars: A Randomized Controlled Trial. J Endod. 2017 Dec;43(12):1953-1962. doi: 10.1016/j.joen.2017.08.007. Epub 2017 Oct 20. PMID 29061359
- [Background] Haak R, Hahnel M, Schneider H, Rosolowski M, Park KJ, Ziebolz D, Hafer M. Clinical and OCT outcomes of a universal adhesive in a randomized clinical trial after 12 months. J Dent. 2019 Nov;90:103200. doi: 10.1016/j.jdent.2019.103200. Epub 2019 Sep 25. PMID 31562889
- [Background] Lawson NC, Robles A, Fu CC, Lin CP, Sawlani K, Burgess JO. Two-year clinical trial of a universal adhesive in total-etch and self-etch mode in non-carious cervical lesions. J Dent. 2015 Oct;43(10):1229-34. doi: 10.1016/j.jdent.2015.07.009. Epub 2015 Jul 29. PMID 26231300
- [Background] Linsuwanont P, Wimonsutthikul K, Pothimoke U, Santiwong B. Treatment Outcomes of Mineral Trioxide Aggregate Pulpotomy in Vital Permanent Teeth with Carious Pulp Exposure: The Retrospective Study. J Endod. 2017 Feb;43(2):225-230. doi: 10.1016/j.joen.2016.10.027. Epub 2016 Dec 29. PMID 28041685
- [Background] Orstavik D, Kerekes K, Eriksen HM. The periapical index: a scoring system for radiographic assessment of apical periodontitis. Endod Dent Traumatol. 1986 Feb;2(1):20-34. doi: 10.1111/j.1600-9657.1986.tb00119.x. No abstract available. PMID 3457698
- [Background] Taha NA, Abdelkhader SZ. Outcome of full pulpotomy using Biodentine in adult patients with symptoms indicative of irreversible pulpitis. Int Endod J. 2018 Aug;51(8):819-828. doi: 10.1111/iej.12903. Epub 2018 Feb 27. PMID 29397003
- [Background] Taha NA, Khazali MA. Partial Pulpotomy in Mature Permanent Teeth with Clinical Signs Indicative of Irreversible Pulpitis: A Randomized Clinical Trial. J Endod. 2017 Sep;43(9):1417-1421. doi: 10.1016/j.joen.2017.03.033. Epub 2017 Jun 30. PMID 28673494
- [Background] Uesrichai N, Nirunsittirat A, Chuveera P, Srisuwan T, Sastraruji T, Chompu-Inwai P. Partial pulpotomy with two bioactive cements in permanent teeth of 6- to 18-year-old patients with signs and symptoms indicative of irreversible pulpitis: a noninferiority randomized controlled trial. Int Endod J. 2019 Jun;52(6):749-759. doi: 10.1111/iej.13071. Epub 2019 Jan 30. PMID 30638262
- [Background] Wolters WJ, Duncan HF, Tomson PL, Karim IE, McKenna G, Dorri M, Stangvaltaite L, van der Sluis LWM. Minimally invasive endodontics: a new diagnostic system for assessing pulpitis and subsequent treatment needs. Int Endod J. 2017 Sep;50(9):825-829. doi: 10.1111/iej.12793. No abstract available. PMID 28776717